CLINICAL TRIAL: NCT01547676
Title: Prospective Randomized Comparison of Clamped Versus Unclamped Partial Nephrectomy
Brief Title: Clamped or Unclamped Surgery in Treating Patients With Kidney Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: P.I. decided to terminate study due to multiple unresolved issues
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4K-10-2; NCI-2012-00057 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-10; First posted 2012-03-08 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Recurrent Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (unclamped partial nephrectomy) (Experimental): Patients undergo unclamped partial nephrectomy. Some patients may undergo unclamped partial nephrectomy with controlled hypotension.
  Interventions: Procedure: robot-assisted laparoscopic surgery
- Arm B (clamped partial nephrectomy) (Active Comparator): Patients undergo clamped partial nephrectomy.
  Interventions: Procedure: robot-assisted laparoscopic surgery

INTERVENTIONS:
Procedure: robot-assisted laparoscopic surgery — Unclamped partial nephrectomy
  Arms: Arm A (unclamped partial nephrectomy)
Procedure: robot-assisted laparoscopic surgery — Undergo clamped partial nephrectomy
  Arms: Arm B (clamped partial nephrectomy)

SUMMARY:
This randomized pilot trial studies clamped or unclamped surgery in treating patients with kidney cancer. Unclamped surgery for kidney cancer may have fewer side effects

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To compare the changes in renal function (post-operative compared to pre-operative) in patients undergoing unclamped partial nephrectomy with or without controlled hypotension (Arm A) vs. those undergoing partial nephrectomy with hilar clamping (Arm B), as measured by change in estimated glomerular filtration rate (eGFR). SECONDARY OBJECTIVES: I. To compare the changes in renal function (post-operative compared to pre-operative) in patients undergoing unclamped partial nephrectomy with or without controlled hypotension (Arm A) vs. those undergoing partial nephrectomy with hilar clamping (Arm B), as measured by change in MAG3 (% of function attributed to affected kidney) and change in serum creatinine. II. To evaluate the safety of the unclamped procedure by estimating the differences in complication rates in patients undergoing unclamped partial nephrectomy with or without controlled hypotension (Arm A) vs. patients undergoing partial nephrectomy with hilar clamping (Arm B) in terms of intra-operative complications and post-operative complications. III. To evaluate the surgical effectiveness of the unclamped procedure by estimating the differences between patients undergoing unclamped partial nephrectomy with or without controlled hypotension (Arm A) vs. patients undergoing partial nephrectomy with hilar clamping (Arm B) in terms of surgical margin status, estimated blood loss, and transfusion rate (intraoperative and post-operative). TERTIARY OBJECTIVES: I. To record and compare the intrarenal blood flow and resistive index measurements in order to determine if a relationship exists between intraoperative findings and postoperative renal function. II. To quantify the amount of acute kidney injury (AKI) and compare the differences between patients undergoing unclamped partial nephrectomy with or without controlled hypotension (Arm A) vs. patients undergoing partial nephrectomy with hilar clamping (Arm B) as measured by urinary and serum biomarkers. III. To compare the effects of the unclamped procedure (Arm A) to the clamped procedure (Arm B) in patients with baseline eGFR < 60, and in patients with age >= 75 (exploratory subset analyses). OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM A: Patients undergo unclamped partial nephrectomy. Some patients may undergo unclamped partial nephrectomy with controlled hypotension. ARM B: Patients undergo clamped partial nephrectomy. After completion of study treatment, patients are followed up at 1 week and then at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Solitary renal mass or solitary complex renal cyst Bosniak >/= Grade 3
* Clinical stage T1a, T1b
* Body Mass Index (BMI) < 40
* Surgical candidate (preoperative cardiac and anesthesia clearance obtained)
* Able to give informed consent
* 24 hour urine collection complete and report obtained
* MAG-3/DTPA scan completed and report obtained

Exclusion Criteria:

* Pregnancy
* More than 1 renal mass or complex renal cyst Bosniak >/= Grade 3 on ipsilateral kidney
* Previous renal surgery on the ipsilateral kidney
* Clinical Stage T2 or greater
* BMI > 40
* Contraindication to systemic hypotension:

  * Left Main Coronary Arterial Disease
  * Severe cardiac decompensation (ejection fraction [EF] < 40%)
  * Prior history of cerebrovascular accident
* Unable to consent
* Unwilling or unable to potentially receive blood transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-12; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in renal function as measured by eGFR | Up to 1 year
  Measured by eGFR, MAG-3 Nuclear Renal Scan, and serum creatinine. The two arms will be compared using regression methods that will account for repeated measures and the pre-randomization stratification.

SECONDARY OUTCOMES:
Estimated blood loss during surgery | Up to 1 year
Rate of blood transfusion during and after surgery | Up to 1 year
Number of patients with positive surgical margins | Up to 1 year
Number of patients with complications during surgery and at 90 days post surgery | Up to 1 year
Number of patients with adverse events | Up to 1 year
Intra-renal blood flow measurements | Up to 1 year
Resistive index measurements | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Desai, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States